CLINICAL TRIAL: NCT03323411
Title: Community-based End-of-Life Intervention for African American Dementia Caregivers
Brief Title: End-of-life Intervention for African American Dementia Caregivers
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Gloria J. Bonner, Principal Investigator, University of Illinois at Chicago
Other Study IDs: 2013-0494; 5R01AG043485-05 (NIH)
Record Dates: First submitted 2017-10-05; First posted 2017-10-27 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Encephalopathy, Ischemic
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention and attention control: the Advance Care Treatment Plan experimental group received education on dementia cardiopulmonary resuscitation and tube feeding. The attention control group received education on exercise stress control diabetes and hypertension
  Interventions: Behavioral: Advance Care Treatment Plan

INTERVENTIONS:
Behavioral: Advance Care Treatment Plan — subjects in experimental group are taught information on dementia mechanical ventilation tube feeding and cardiopulmonary resuscitation

SUMMARY:
In a community-based approach, the investigators long-term goal is to empower African American family caregivers who are designated healthcare proxies to make informed end-of-life treatment decisions for participants with moderate to severe dementia before a life-threatening medical crisis occurs.

DETAILED DESCRIPTION:
The investigators conducted a randomized controlled trial for efficacy of the Advance Care Treatment Program in an African American church-based community model. The investigators compared the effect of the experimental and control groups on knowledge, self-efficacy, intentions and behaviors from 4 urban African American churches randomly assigned to experimental (n=2) or control (n=2) conditions,304 (experimental n=152; control (n=152) health care proxies of participants that have advanced stage dementia: (a) were concurrently recruited in small classes each with 8-9 healthcare proxies.

ELIGIBILITY:
"Inclusion Criteria"

* Caregiver spouse or adult child of care recipient
* Caregiver knowledgeable about care recipient's medical history
* Care recipient must be African American
* Care recipient must have moderate to severe stage dementia
* Care recipient must lack decisional capacity

"Exclusion Criteria"

* Not a caregiver
* Care recipient not African American,
* Care recipient without moderate to severe dementia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — 301 african american females and 54 african american males
Study Population: African American family caregivers over the age of 18 who attend four specific urban mega churches who meet the eligibility criteria for the study.
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2013-08-15 (Actual); Primary Completion 2016-09-10 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Knowledge of dementia | Three years
  Knowledge of Dementia Scale measures Knowledge of dementia with 17 dichotomous true/false items, maximum total score = 17 and Cronbach's α=.76. Higher scores indicate greater practical understanding of dementia knowledge
Knowledge of cardiopulmonary resuscitation (CPR), mechanical ventilation (MV), tube feeding (TF) | Three years
  Knowledge of CPR, MV, and TF Scale mmeasures CPR, MV and TF with 18-items Likert (5-point) and yes/no questions. Higher scores indicate increased general knowledge of CPR, MV and TF.
Self efficacy | Three years
  Confidence in Treatment Decisions Made Scale measures self-efficacy on decision choices for CPR, MV, and TF with12-item Likert scale (1=extremely comfortable to 5=not at all comfortable) and Cronbach α=.93
Intention to make a Care Plan | Three years
  Treatment Decisions Questionnaire measured Intention to make a Care Plan using the 3-item dichotomous (yes/no) items on each CPR, MV and TF.

SECONDARY OUTCOMES:
Written Care Plan | 3 years
  Treatment Decision Questionnaire 3 items dichotomous yes/no measuring actual care plan implemented on CPR, MV, TF

CONTACTS AND LOCATIONS:
Overall Officials: Gloria J Bonner, PhD, Principal Investigator — University of Illinois at Chicago

IPD SHARING:
Plan to Share IPD: No